CLINICAL TRIAL: NCT05956613
Title: Evaluation of Postoperative Pain After Partial Pulpotomy Versus Full Root Canal Treatment in Managing Young Permanent Molars With Symptomatic Irreversible Pulpitis: a Randomized Controlled Trial
Brief Title: Post Operative Pain of Partial Pulpotomy Using a Bioceramic Material in Patients With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Omaia Ahmed Salah, Lecturer of Endodontics, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECO6U/27-2023
Record Dates: First submitted 2023-07-07; First posted 2023-07-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Endodontic Disease
Keywords: bioceramic material, pulpitis, partial pulpotomy
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: conventional root canal treatment (No Intervention)
- Test: partial pulpotomy (Other): Partial pulpotomy using bioceramic putty
  Interventions: Procedure: Partial pulpotomy

INTERVENTIONS:
Procedure: Partial pulpotomy — Use of newly introduced bioceramic putty in partial pulpotomy
  Arms: Test: partial pulpotomy

SUMMARY:
The goal of this clinical trial is to assess post-operative pain of partial pulpotomy using a newly introduced Bioceramic material in young patients with symptomatic irreversible pulpitis at 24, 48, 72 hours postoperatively using visual analogue scale (VAS). The main question[s] it aims to answer are:

• In patients with symptomatic irreversible pulpitis does the use of bioceramic material in partial pulpotomy decrease amount of post operative pain in comparison to conventional root canal treatment?

Participants will record the intensity of pain at 24,48, 72 hours postoperatively.

ELIGIBILITY:
1. Inclusion criteria :

   1. Subject's age between 9-14 years.
   2. Both male and female subjects.
   3. Medically free and healthy subjects.
   4. Mandibular molar teeth.
   5. Teeth with symptomatic irreversible pulpitis.
   6. Teeth with mature closed apices.
2. Exclusion Criteria:

   1. Teeth with acute dentoalveolar abscess.
   2. Subjects having more than one tooth that require root canal treatment.
   3. Subjects that have taken analgesic, anti-inflammatory or antibiotic drugs during the 10 days prior to the start of treatment.
   4. Subjects with systemic diseases who have endocrine diseases, Infectious diseases or Psychological disturbance.
   5. Teeth with periodontal disease or pulp calcification.
   6. Subjects taking chronic pain medications.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Post operative pain | after 24 hours
  Measure intensity of post operative pain using visual analogue scale (VAS)
Post operative pain | after 48 hours
  Measure intensity of post operative pain using visual analogue scale (VAS)
Post operative pain | After 72 hours
  Measure intensity of post operative pain using visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No